CLINICAL TRIAL: NCT06943846
Title: Wound Healing Outcomes in Aged Extraction Patient With Platelet Rich Fibrinogen
Brief Title: Platelet-Rich Fibrinogen in Extraction Socket Healing of the Aged
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 0153-25-FB
Record Dates: First submitted 2025-03-18; First posted 2025-04-24 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Edentulism
Keywords: extraction; platelet-rich; fibrin; healing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aged Participants Treated with Platelet-rich Fibrinogen (Active Comparator): Participants aged 50 to 80 years of age will receive Platelet-rich Fibrinogen (PRF) treatment after tooth extraction.
  Interventions: Procedure: Platelet-rich fibrin (PRF)
- Aged Control (No Intervention): Participants aged 50 to 80 years of age will not receive Platelet-rich Fibrinogen (PRF) treatment after tooth extraction.
- Young Participants Treated with Platelet-rich Fibrinogen (Active Comparator): Participants aged 14 to 18 years of age will receive Platelet-rich Fibrinogen (PRF) treatment after tooth extraction.
  Interventions: Procedure: Platelet-rich fibrin (PRF)
- Young Control (No Intervention): Participants aged 14 to 18 years of age will not receive Platelet-rich Fibrinogen (PRF) treatment after tooth extraction.

INTERVENTIONS:
Procedure: Platelet-rich fibrin (PRF) — Platelet-rich fibrin added to extraction socket
  Arms: Aged Participants Treated with Platelet-rich Fibrinogen; Young Participants Treated with Platelet-rich Fibrinogen

SUMMARY:
The purpose of this study is to better understand oral wound healing in the aged participant following placement of platelet-rich fibrinogen (PRF). In this study, 12 participants requiring a posterior tooth extraction will be enroll: 6 participants aged 14-18, 6 participants aged 50-80. All will undergo a posterior tooth extraction with a small tissue specimen taken from the extraction site. Half of the participants will also have their blood drawn and platelet-rich fibrinogen placed in the extraction socket. Participants will return in 2 weeks for suture removal and another soft tissue sample. Participants will return at 3 months for a final post-operative radiograph. All soft tissue samples will undergo immunofluorescence.

DETAILED DESCRIPTION:
Twelve participants who are patients at the University of Nebraska Medical Center College of Dentistry who are seeking care to extract a posterior tooth (premolar, molar) due to a periodontal or endodontic defect, non-restorable caries or fracture, serial extractions for orthodontic purposes and who are considering a dental implant to replace the extracted tooth, will be enrolled. On the day of extraction, baseline data will be collected: gender, smoking status and medical history. Hemoglobin A1C (HbA1C) will be tested via a simple finger prick to determine if participant's long-term blood glucose levels could be associated to oral wound healing. A peripheral blood draw will be obtained for platelet-rich fibrinogen (PRF) application.

Prior to extraction, clinical measurements [probing depth (PD), recession, and bleeding on probing (BOP)] will be collected at 6 sites (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, distolingual) to assess inflammatory periodontitis severity. A limited-field cone beam commuted tomography (CBCT) radiograph will be taken to assess bone anatomy for future extraction/implant planning and to confirm the probable lack of need for bone augmentation/grafting following extraction. Gingival crevicular fluid (GCF) will be sampled at the interproximal sites of teeth adjacent to the tooth to be extracted. The tooth to be extracted will be isolated with cotton rolls and gingival crevicular fluid (GCF) collection paper strips will be placed into the facial and lingual interproximal gingival sulci for 30 seconds. The paper samples will be pooled and placed in a plastic-capped vial labeled with the participant's number and visit and immediately frozen at -80° C. The presence of explorer-detectable plaque will be ascertained on 6 sites (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, distolingual) on tooth to be extracted and adjacent teeth.

Routine atraumatic dental extraction under local anesthesia will be completed by the assigned periodontal resident and faculty. Immediately after the extraction, the resident/fellow will remove a small piece of gingival/mucosal tissue (approximately 3 mm x 3 mm x 3 mm) from the mesial or distal interproximal sites of the extracted tooth and suture the site with chromic gut suture. Soft tissue samples will be immediately placed in formalin. Participants will be scheduled for a routine post-operative visit one, two or three weeks following the extraction. At this visit, suture removal and evaluation of healing site will occur. GCF collection on the remaining adjacent teeth will occur as will collection of granulation tissue (3 mm x 3 mm x 3 mm) from the extraction site. Due to minimal/lack of innervation of granulation tissue, it is not anticipated that anesthesia will be necessary to collect a sample, however, local anesthesia can be administered if the participant reports sensitivity at suture removal. The final post-operative visit will be 3 months following the extraction. A limited-field cone-beam computed tomography (CBCT) will be taken to begin the process of implant treatment planning for bone height, width and volume. All baseline clinical measures (PD/recession/BOP) as well as GCF sampling will be completed on adjacent teeth. The soft tissue samples will be processed for immunofluorescence.

ELIGIBILITY:
Inclusion Criteria:

* Patient at University of Nebraska Medical Center (UNMC) College of Dentistry
* Requires extraction of posterior tooth
* Able and willing to provide consent/assent

Exclusion Criteria:

* Systemic conditions that delay wound healing
* Chronic use of non-steroidal anti-inflammatory drugs (NSAIDs), methotrexate, bisphosphonates or other drugs that inhibit wound healing Smoking and vaping Pregnancy

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Cytokine Concentration | Baseline and two weeks post-extraction
  Indirect immunofluorescent intensity will determine concentration of cytokines present in sample.

SECONDARY OUTCOMES:
Bone Density | 3 months post-extraction
  Bone density as measured through cone beam computed tomography (CBCT) and Hounsfeld units will determine density of new bone formation.

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Killeen, DDS, MS, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center College of Dentistry, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No